CLINICAL TRIAL: NCT01581814
Title: Effects of Drospirenone-ethinylestradiol and/or Metformin on Cardiovascular Risk in Hyperinsulinemic Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: disfunzionale14
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin (Active Comparator): 31 subjects were randomized to receive 500 mg Metformin per 3/die
  Interventions: Drug: Metformin
- 0.03 mg EE plus 3 mg of DRPS (Active Comparator)
  Interventions: Drug: Yasmin;
- Metformin plus Yasmin (Active Comparator)
  Interventions: Drug: Metformin plus Yasmin

INTERVENTIONS:
Drug: Metformin — 500 mg of Metformin per 3/die
  Arms: Metformin
Drug: Yasmin; — 1pill/day for cycles of 28 days (21 pills followed by 7 no-pill days)
  Arms: 0.03 mg EE plus 3 mg of DRPS
Drug: Metformin plus Yasmin — 0.03 mg EE plus 3 mg of DRPS combined with 500 mg of metformin three times daily
  Arms: Metformin plus Yasmin

SUMMARY:
To evaluate long-term effects of drospirenone (DRSP)/ethinylestradiol (EE) alone, metformin alone and DRSP/EE plus metformin on some cardiovascular risk factors in hyperinsulinemic PCOS patients

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS), one of the most common endocrine disorders affecting women on reproductive age , seems to be associated with an increased incidence of cardiovascular disease. At present, insulin-sensitizing drugs, such as metformin, represent one of the most important line treatment for hyperinsulinemic PCOS women. Metformin is able to produce favourable outcomes on the metabolic derangements in insulin-resistant normal weight and obese PCOS patients. Oral contraceptives represent the traditional medical therapy for the long-term treatment of PCOS women, in order to obtain regular menstrual cycles and to improve the clinical signs of hyperandrogenism.Based on the above mentioned evidences, the aim of the present study was to evaluate the effects of DRPS/EE alone versus metformin alone versus DRPS/EE plus metformin on the CD4+CD28null T cells frequency and on endocrino-metabolic parameters, in hyperinsulinemic PCOS patients

ELIGIBILITY:
Inclusion Criteria:

* age 18-35
* hyperinsulinemic PCOS

Exclusion Criteria:

* chronic or acute inflammatory disease, cancer, autoimmune disease, treatment with clomiphene citrate, oral contraceptives, antiandrogens, drugs to control appetite or insulin-sensitizing drugs (metformin, pioglitazone and rosiglitazone) during the last 6 months prior to our evaluation, DM2, hypertension, major surgery in the last 3 months or other hormonal dysfunctions (hypothalamic, pituitary, thyroidal, or adrenal causes).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
CD4+CD28null frequency | five minutes

SECONDARY OUTCOMES:
the area under the curve for insulin (AUCi) and lipid profile. | 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico A. Gemelli, Rome, Rome, Italy

REFERENCES:
- [Result] Niccoli G, Apa R, Lanzone A, Liuzzo G, Spaziani C, Sagnella F, Cosentino N, Moro F, Martinez D, Morciano A, Baca M, Pazzano V, Gangale MF, Tropea A, Crea F. CD4+CD28 null T lymphocytes are expanded in young women with polycystic ovary syndrome. Fertil Steril. 2011 Jun 30;95(8):2651-4. doi: 10.1016/j.fertnstert.2011.01.129. Epub 2011 Feb 16. PMID 21324454